CLINICAL TRIAL: NCT03854383
Title: Efficacy of Intravaginal Administration of Isosorbide Mononitrate Together With Misoprostol Versus Misoprostol Alone in Induction of Labor in Postdate Women
Brief Title: Using Isosorbide Mononitrate in Reducing Time in Induction of Labor in Post Date Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abdelrahman Ali Fadel Youssef Mohamed (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Ali Fadel Youssef Mohamed, Principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 600181
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Induction of Labor
MeSH Terms: interventions — isosorbide-5-mononitrate; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol alone (Sham Comparator): Enrolled women will receive 25 πg of misoprostol which will be placed intravaginally 4 hourly, maximum up to 5 doses
  Interventions: Drug: Misoprostol
- Isosorbide mononitrate with misoprostol (Active Comparator): Enrolled women will receive 25 πg of misoprostol together with 40 mg isosorbide mononitrate which will be placed intravaginally 4 hourly, maximum up to 5 doses
  Interventions: Drug: Isosorbide mononitrate; Drug: Misoprostol

INTERVENTIONS:
Drug: Isosorbide mononitrate — Administration of isosorbide mononitrate vaginaly together with misoprostol in induction of labor in postdate women
  Arms: Isosorbide mononitrate with misoprostol
Drug: Misoprostol — Used intravaginally to ripe the cevix in induction of labor

SUMMARY:
We will compare between using isosorbide mononitrate together with misoprostol versus the misoprostol alone in induction of labor in postdate women

ELIGIBILITY:
Inclusion Criteria:

* age (20-35 yrs)
* single fetus
* gestational age > 40weeks
* not in labor
* bishop score < 7
* no medical disorder

Exclusion Criteria:

* Gestational age ≤40 weeks
* patient with a ripe cervix
* rupture of membranes
* suspected chorioamnionitis
* placenta previa
* history of major uterine surgery
* hypertonic uterine pattern
* contraindicated to receive PG
* fetal malpresentation
* multiple pregnancy
* intrauterine growth retardation
* women with any general medical disorder

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-03 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
The duration of induction to active phase interval | 12 weeks
  Measure the time between the beginning of the induction to enter the active phase of labor

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt